CLINICAL TRIAL: NCT06518616
Title: Reducing Psychological Distress in Fire Fighters With an Asynchronous App- Based Meditation Intervention
Brief Title: Meditation to Reduce Firefighter Distress
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003422
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Psychological Distress

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-day meditation intervention (Experimental): prerecorded meditation units, 10 units, one per day, delivered by smartphone app
  Interventions: Behavioral: 10-day meditation intervention
- 10-day health education intervention (Active Comparator): prerecorded health education units, 10 units, one per day, delivered by smartphone app
  Interventions: Behavioral: 10-day health education intervention

INTERVENTIONS:
Behavioral: 10-day meditation intervention — prerecorded meditation units delivered by smartphone app
  Arms: 10-day meditation intervention
Behavioral: 10-day health education intervention — prerecorded health education units delivered by smartphone app
  Arms: 10-day health education intervention

SUMMARY:
The more than one million firefighters in the United States provide critical emergency medical services in communities they serve and are on the front lines of healthcare delivery, including in the post-pandemic world. As a result of exposure to occupational stressors, a high proportion of firefighters experience considerable stress-related burden including psychological distress (i.e., increased features of anxiety and depression). To address this need, this project will test the efficacy of a 10-day meditation intervention (i.e., 10 individual prerecorded audio units delivered by smartphone app) among career firefighters to decrease psychological distress (i.e., anxiety and depression).

DETAILED DESCRIPTION:
The goal of this study is to test the efficacy of a 10-day meditation intervention (i.e., 10 individual prerecorded audio units delivered by smartphone app) versus an active attention control (i.e., 10-day health education intervention with 10 individual prerecorded audio units delivered by smartphone app) to reduce psychological distress among N=160 career firefighters (to address possible attrition, N=192 firefighters will be consented and enrolled). The following specific aims will guide the research:

Aim 1. Examine whether firefighters' psychological distress (i.e., features of anxiety [primary outcome], depression) is reduced at 10 days, 30 days, and 3 months after the meditation intervention versus an active attention control. Features of anxiety, features of depression will be assessed at baseline (T1), after the 10-day intervention (T2), 30 days later (T3), and 3 months later (T4).

Aim 2: Explore the extent to which reductions in psychological distress from the meditation intervention are mediated by mindfulness and perceived social connection.

ELIGIBILITY:
Inclusion criteria: 1) currently employed as a career firefighter, 2) 18 or older, 3) speak and understand English, and 4) own a smartphone (iPhone or Android) able to download and run the intervention apps.

Exclusionary factors: 1) diagnosis of an illness requiring use of corticosteroids (e.g., asthma), and 2) have ongoing or past regular meditation experience in the last 4 years (i.e. more than two meditation session [completed or attempted] per year either with a group or individually), as determined by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
anxiety features | before, immediately after, 30 days after, and 3 months after the 10-day interventions
  PROMIS (Patient Reported Outcomes Measurement Information System) Short Form Emotional Distress - Anxiety - 8a

SECONDARY OUTCOMES:
depression features | before, immediately after, 30 days after, and 3 months after the 10-day interventions
  PROMIS Short Form Emotional Distress - Depression - 8a

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus Pace, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No